CLINICAL TRIAL: NCT06343376
Title: A Phase I Trial of CD19-Targeted Chimeric Antigen Receptor (CAR) Modified T Cells Genetically Engineered to Secrete Interleukin 12 (IL-12) and With a Truncated Human Epidermal Growth Factor Receptor (EGFRt) in Patients With Relapsed or Refractory CD19+ Hematologic Malignancies
Brief Title: Genetically Engineered Cells (EGFRt/19-28z/IL-12 CAR T Cells) for the Treatment of Relapsed or Refractory CD19+ Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Manufacturing issues
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-3641523; NCI-2024-01818 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3641523 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-03-25; First posted 2024-04-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Transformed Chronic Lymphocytic Leukemia; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Transformed Chronic Lymphocytic Leukemia; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Biopsy; Specimen Handling; Cyclophosphamide; fludarabine phosphate; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (EGFRt/19- 28z/IL-12 CAR T cells) (Experimental): Patients undergo leukapheresis prior to treatment. Patients receive EGFRt/19- 28z/IL-12 CAR T cells IV over 5 to 30 minutes on day 0. Patients also undergo ECHO or MUGA during screening. Patients also undergo CT or PET as well as bone marrow biopsy and aspiration and blood sample collection throughout the trial. Additionally, patients undergo a tissue biopsy during screening and on the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography; Biological: EGFRt/19-28z/IL-12 CAR T-lymphocytes; Procedure: Leukapheresis; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography
- Cohort B (EGFRt/19- 28z/IL-12 CAR T cells, conditioning) (Experimental): Patients undergo leukapheresis prior to treatment and receive lymphodepletion chemotherapy with cyclophosphamide IV over 2 hours and fludarabine IV over 30 minutes on days -5, -4, and -3. Patients then receive EGFRt/19- 28z/IL-12 CAR T cells IV over 5 to 30 minutes on day 0. Patients also undergo ECHO or MUGA during screening. Patients also undergo CT or PET as well as bone marrow biopsy and aspiration and blood sample collection throughout the trial. Additionally, patients undergo a tissue biopsy during screening and on the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Biological: EGFRt/19-28z/IL-12 CAR T-lymphocytes; Drug: Fludarabine Phosphate; Procedure: Leukapheresis; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
  Arms: Cohort B (EGFRt/19- 28z/IL-12 CAR T cells, conditioning)
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Biological: EGFRt/19-28z/IL-12 CAR T-lymphocytes — Given IV
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
  Arms: Cohort B (EGFRt/19- 28z/IL-12 CAR T cells, conditioning)
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of genetically engineered cells called EGFRt/19-28z/IL-12 CAR T cells, and to see how they work in treating patients with hematologic malignancies that makes a protein called CD19 (CD19-positive) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Chimeric Antigen Receptor (CAR) T-cell Therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. To improve the effectiveness of the modified T cells and to help the immune system fight cancer cells better, the modified T cells given in this study will include a gene that makes the T cells produce a cytokine (a molecule involved in signaling within the immune system) called interleukin-12 (IL-12). The researchers think that IL-12 may improve the effectiveness of the modified T cells, and it may also strengthen the immune system to fight cancer. Giving EGFRt/19-28z/IL-12 CAR T cells may be safe and tolerable in treating patients with relapsed or refractory CD19+ hematologic malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, toxicity and maximum tolerated dose (MTD) of EGFRt/19-28z/IL-12 CAR T-lymphocytes (EGFRt/19-28z/IL-12 CAR T cells) in patients with relapsed or refractory CD19+ aggressive hematologic malignancies.

SECONDARY OBJECTIVES:

I. To assess the anti-tumor efficacy of adoptively transferred EGFRt/19-28z/IL-12 T cells.

II. To assess the in vivo persistence of adoptively transferred EGFRt/19-28z/IL-12 T cells.

EXPLORATORY OBJECTIVES:

I. To describe the cellular and cytokine microenvironment following infusion of adoptively transferred EGFRt/19-28z/IL-12 T cells.

II. To characterize endogenous anti-tumor immune responses following infusion of adoptively transferred EGFRt/19-28z/IL-12 T cells.

III. To summarize levels of normal B cells and the incidence of B cell aplasia following infusion of adoptively transferred EGFRt/19-28z/IL-12 T cells.

IV. To determine the proportion of evaluable patients who achieve minimal residual disease (MRD)-negativity in peripheral blood and/or bone marrow.

V. To assess phenotype and in vitro function of end-of-production (EOP) EGFRt/19-28z/IL-12 CAR T cells and phenotype at recovery following CAR T cell administration.

OUTLINE: This is a dose-escalation study of EGFRt/19- 28z/IL-12 CAR T cells. Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients undergo leukapheresis prior to treatment. Patients receive EGFRt/19- 28z/IL-12 CAR T cells intravenously (IV) over 5 to 30 minutes on day 0. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients also undergo computed tomography (CT) or positron emission tomography (PET) as well as bone marrow biopsy and aspiration and blood sample collection throughout the trial. Additionally, patients undergo a tissue biopsy during screening and on the trial.

COHORT B: Patients undergo leukapheresis prior to treatment and receive lymphodepletion chemotherapy with cyclophosphamide IV over 2 hours and fludarabine IV over 30 minutes on days -5, -4, and -3. Patients then receive EGFRt/19- 28z/IL-12 CAR T cells IV over 5 to 30 minutes on day 0. Patients also undergo ECHO or MUGA during screening. Patients also undergo CT or PET as well as bone marrow biopsy and aspiration and blood sample collection throughout the trial. Additionally, patients undergo a tissue biopsy during screening and on the trial.

After completion of study treatment, patients are followed up weekly for 4 weeks, every 4 weeks until 24 months, every 3 months thereafter for 1 year, then annually for up to 5 years, followed by long-term follow up for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed refractory B Cell malignancies which commonly express CD-19.

  * Eligible disease subtypes include the following:

    * Patients with diffuse large B-cell lymphoma (de novo or diffuse large B-cell lymphoma [DLBCL] transformed from an indolent lymphoma (follicular lymphoma, chronic lymphocytic leukemia) or high grade B-cell Lymphoma (HGBL):

      * Relapsed or refractory DLBCL or high-grade B-cell lymphoma (HGBL) following 2 or more prior chemoimmunotherapy regimens containing an anthracycline and CD20-directed therapy following diagnosis of de novo DLBCL/HGBL or DLBCL arising from indolent lymphoma and requiring further treatment.
      * Relapse following a single prior chemoimmunotherapy regimen containing an anthracycline and CD20-directed therapy following diagnosis of de novo DLBCL/HGBL or DLBCL arising from indolent lymphoma and considered ineligible for high dose chemotherapy and autologous stem cell rescue as determined by the investigator.
      * Patients must have at least one fludeoxyglucose F-18 (FDG)-avid (PET-avid) measurable lesion.
      * Biopsy confirmation of relapsed or refractory DLBCL is required.
    * Chronic lymphocytic leukemia after 2 lines of therapy including a BTKi (bruton tyrosine kinase inhibitor).
    * Mantle cell lymphoma after 2 lines of therapy. Patients must have previously received chemoimmunotherapy and a prior BTK inhibitor.
    * Follicular lymphoma after 2 lines of therapy.
* For cohort 1A specifically, patients must additionally have received a prior CD19-targeted CAR T-cell therapy or not have an indication for a Food and Drug Administration (FDA)-approved commercial CD19-targeted CAR T-cell therapy. This will include patients with relapsed/refractory DLBCL, FL, CLL and MCL.
* For cohorts other than cohort 1A (and if needed, cohort -1), patients with an indication for an FDA approved commercial CD19-targeted CAR T-cell therapy are eligible following an informed consent discussion that reviews the risks and benefits of the FDA-approved commercial CD19-targeted CAR T-cell therapy vs the investigational product.
* Prior CD19-targeted therapies, including CAR T-cell therapy, does not exclude participation; however, CD19 expression by immunohistochemical staining or flow cytometry must be confirmed prior to enrollment for patients who have received such therapies.
* Age ≥ 18 years of age.
* Creatinine Clearance > 30 mL/min (Cockroft-Gault equation).
* Direct bilirubin ≤ 2.0 mg/dL (unless related to disease).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) (unless related to disease).
* Adequate pulmonary function as assessed by ≥ 90% oxygen saturation on room air by pulse oximetry.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Patients of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Pregnant or lactating patients.
* Impaired cardiac function (left ventricular ejection fraction [LVEF] < 40%) as assessed by ECHO or MUGA scan during screening.
* Patients with active graft versus host disease following allogeneic hematopoietic cell transplantation requiring systemic T cell suppressive therapy are ineligible.
* Patients with active autoimmune disease requiring systemic T cell suppressive therapy are ineligible.
* Patients with following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure.
  * Myocardial infarction ≤ 6 months prior to enrollment.
  * Any history of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration.
* Patients with HIV are ineligible.
* Patients with active hepatitis B infection (as manifest by either detectable hepatitis B virus deoxyribonucleic acid [DNA] by polymerase chain reaction [PCR] and/or positivity for hepatitis B surface antigen) are ineligible.
* Patients with active hepatitis C infection (as manifest by detectable hepatitis C virus ribonucleic acid [RNA] by PCR) are ineligible. Patients with detectable antibodies to hepatitis C virus will be screened by PCR for evidence of active infection.
* Patients with uncontrolled systemic fungal, bacterial, viral or other infection are ineligible.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of skin.
* Patients with history or presence of clinically significant neurological disorders such as epilepsy, generalized seizure disorder, severe brain injuries are ineligible.
* Patients with primary central nervous system (CNS) disease are ineligible.
* Unwilling or unable to follow protocol requirements.
* Any other condition/issue which, in the opinion of the treating physician, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Will be graded on a scale of 1 to 5 as described by the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0).
Maximal tolerated dose (MTD) of EGFRt/19-28z/IL-12 chimeric antigen receptor T-cells | Within 30 days from the final infusion of the EGFRt/19-28z/IL-12 T cells
  Will be defined as the highest dose with an observed incidence of dose limiting toxicities in no more than one out of six patients treated at a particular dose level. Will be assessed using NCI CTCAE v 5.0.

SECONDARY OUTCOMES:
Incidence of complete remission (CR)/complete remission with incomplete count recovery (CRi) | Within 3 months of CAR T-cell infusion
Incidence of CR/CRi + partial response (PR) (ORR) | Within 3 months of CAR T-cell infusion
Event free survival | Up to 5 years
  Will be computed using the Kaplan- Meier method.
Overall survival | Up to 5 years
  Will be computed using the Kaplan- Meier method.
Progression-free survival | Up to 5 years
Modified T-cell persistence | Up to 5 years
  Will be determined by the presence of detectable CAR T-cells (quantitative polymerase chain reaction or multiparameter flow cytometry).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Hernandez-ILizaliturri, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States